CLINICAL TRIAL: NCT00178048
Title: Paroxetine in the Treatment of Chronic Primary Insomnia: A Double-Blind, Randomized, Placebo-Controlled Study of Efficacy Over Six Weeks
Brief Title: Paroxetine in the Treatment of Chronic Primary Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 970357
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Primary Insomnia; Depression
Keywords: primary insomnia; insomnia; depression; late life; elderly; sleep disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Sleep Wake Disorders | interventions — Paroxetine

INTERVENTIONS:
Drug: paroxetine

SUMMARY:
The goal of the study is to examine the role of paroxetine, an antidepressant medication, in the acute and continuation treatment of insomnia. Primary insomnia is a type of insomnia not directly resulting from general medical, chemical, or psychiatric conditions.

DETAILED DESCRIPTION:
The primary aim of this study is to demonstrate the role of paroxetine in the acute treatment of chronic primary insomnia. Paroxetine taken on a nightly basis in combination with sleep hygiene therapy will produce a greater number of diagnostic responders in acute treatment, compared to a placebo and sleep hygiene control condition, in a randomized, double-blinded, six-week acute treatment trial. EEG sleep, sleep quality, and daytime well-being, and daytime functioning will also show superior treatment effects during acute treatment with paroxetine plus sleep hygiene, as compared with the placebo control condition.

A total of 66 patients with primary insomnia, as defined by DSM-IV criteria, will be randomized (1:1) to receive paroxetine plus sleep hygiene therapy (P+SH-a) or placebo plus sleep hygiene therapy (PL+SH-a) in weekly acute treatment sessions evolving over a six-week interval in a double-blinded, parallel group design.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 or older
* Diagnosis of chronic primary insomnia
* Score of 8 or higher on the Pittsburgh Sleep Quality Index
* free of all antidepressants and benzodiazepine for two weeks

Exclusion Criteria:

* lifetime diagnosis of any psychotic disorder,or bipolar disorder.
* DSM-IV diagnosis of dysthymia or generalized anxiety disorder
* Diagnosis of major depression within the past 6 months
* Alcohol or drug abuse within the past 6 months
* Contraindication to SSRI therapy
* History of seizure disorder
* Baseline apnea/hypopnea index score greater than 15
* Hyponatremia

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66
Dates: Start 1998-09; Study Completion 2003-12

PRIMARY OUTCOMES:
Paroxetine in combination with sleep hygiene therapy will produce a greater number of responders in acute treatment, compared to a placebo and sleep hygiene condition, in a randomized, double-blinded, six-week acute trial

SECONDARY OUTCOMES:
Polysomnographic Sleep measures
Pittsburgh Sleep Quality Index and Sleep Diary
Daytime well being on the Profile of Mood States
Daytime functioning on the Sickness Impact Profile, Medical Outcomes Study (SF-36), and UKU
Stress measures: Schedule of Recent Events, Perceived Stress Scale, Impact of Life Events Scale, Ways of Coping Inventory, Multidimensional Fatigue Inventory, and Brief Symptom Inventory
Psychophysiological arousal and mood measures collected at each sleep study: the Pres-Sleep Arousal Scale, Spielman Insomnia Symptom Questionnaire, Pittsburgh Insomnia Rating Scale, and the Pre-Sleep Experience Questionnaire.
SCID
Sleep Hygiene Awareness and Practices Scale
Diagnostic Response: Clinical Global Impressions Scale

CONTACTS AND LOCATIONS:
Overall Officials: Charles F Reynolds III, M.D., Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Pittsubrgh Medical Center, Pittsburgh, Pennsylvania